CLINICAL TRIAL: NCT02392234
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Crossover Study to Evaluate the Efficacy and Safety of Ivacaftor and VX-661 in Combination With Ivacaftor in Subjects Aged 12 Years and Older With Cystic Fibrosis, Heterozygous for the F508del-CFTR Mutation, and a Second Allele With a CFTR Mutation Predicted to Have Residual Function
Brief Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Ivacaftor and VX-661 in Combination With Ivacaftor in Subjects Aged 12 Years and Older With Cystic Fibrosis, Heterozygous for the F508del-cystic Fibrosis Transmembrane Conductance Regulator (CFTR) Mutation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: VX14-661-108; 2014-004788-18 (EudraCT Number)
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- VX-661/Ivacaftor combination (Experimental)
  Interventions: Drug: VX-661/Ivacaftor; Drug: Ivacaftor; Drug: Placebo matched to Ivacaftor
- Ivacaftor monotherapy (Experimental)
  Interventions: Drug: Ivacaftor; Drug: Placebo matched to VX-661/ ivacaftor
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matched to VX-661/ ivacaftor; Drug: Placebo matched to Ivacaftor

INTERVENTIONS:
Drug: VX-661/Ivacaftor — Fixed dose combination tablet, oral use
  Other Names: VX-661+VX-770
  Arms: VX-661/Ivacaftor combination
Drug: Ivacaftor — Tablet, oral use
  Other Names: IVA, VX-770
  Arms: Ivacaftor monotherapy; VX-661/Ivacaftor combination
Drug: Placebo matched to VX-661/ ivacaftor — Fixed dose combination tablet, oral use
  Arms: Ivacaftor monotherapy; Placebo
Drug: Placebo matched to Ivacaftor — Tablet, oral use
  Arms: Placebo; VX-661/Ivacaftor combination

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of VX-661 in combination with ivacaftor (IVA, VX-770) and IVA monotherapy in participants with Cystic Fibrosis (CF) who are heterozygous for F508del-CFTR allele and a second allele with a CFTR mutation predicted to have residual function.

ELIGIBILITY:
Inclusion Criteria:

* Heterozygous for F508del-CFTR and a second allele with a CFTR mutation predicted to have residual function
* Forced Expiratory Volume in 1 Second (FEV1) greater than or equal to (≥) 40 percent (%) and less than or equal to (≤) 90% of predicted normal for age, sex, and height during screening
* Sweat chloride value ≥60 millimole per liter (mmol/L) during screening OR as documented in the participant's medical record
* Stable CF disease as judged by the investigator

Exclusion Criteria:

* History of any comorbidity that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant
* An acute upper or lower respiratory infection, pulmonary exacerbation
* History of solid organ or hematological transplantation
* Ongoing or prior participation in an investigational drug study (including studies investigating VX-661, lumacaftor [VX-809], and/or ivacaftor) within 30 days of screening
* Pregnant and nursing females
* Sexually active participants of reproductive potential who are not willing to follow the contraception requirements

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2015-03; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (93):
- United States (47):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Long Beach, California
  - Oakland, California
  - Palo Alto, California
  - Sacramento, California
  - Aurora, Colorado
  - Denver, Colorado
  - Gainesville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Park Ridge, Illinois
  - Iowa City, Iowa
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Grand Rapids, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - New York, New York
  - Syracuse, New York
  - Valhalla, New York
  - Chapel Hill, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Sioux Falls, South Dakota
  - Memphis, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Tyler, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Seattle, Washington
  - Spokane, Washington
  - Milwaukee, Wisconsin
- Australia (4):
  - Adelaide
  - Melbourne
  - South Brisbane
  - Westmead
- Ghent, Belgium
- Canada (4):
  - Montreal
  - Québec
  - Toronto
  - Vancouver
- France (7):
  - Marseille, Bouches-du-Rhone
  - Montpellier, Herault
  - Rennes, Ille Et Vilaine
  - Lille, Nord
  - Paris, Paris
  - Bron, Rhone
  - Bordeaux
- Germany (6):
  - Munich, Bavaria
  - München, Bavaria
  - Hanover, Lower Saxony
  - Essen, North Rhine-Westphalia
  - Jena, Thuringia
  - Berlin
- Israel (4):
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
- Italy (6):
  - Ancona
  - Milan
  - Orbassano
  - Potenza
  - Roma
  - Verona
- Netherlands (4):
  - Amsterdam
  - Rotterdam
  - The Hague
  - Utrecht
- Switzerland (3):
  - Bern
  - Sankt Gallen
  - Zurich
- United Kingdom (7):
  - Exeter, Devon
  - London, Greater London
  - Manchester, Greater Manchester
  - Southampton, Hampshire
  - Liverpool, Lancashire
  - Glasgow, Strathclyde
  - Leeds, West Yorkshire

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Acaster S, Mukuria C, Rowen D, Brazier JE, Wainwright CE, Quon BS, Duckers J, Quittner AL, Lou Y, Sosnay PR, McGarry LJ. Development of the Cystic Fibrosis Questionnaire-Revised-8 Dimensions: Estimating Utilities From the Cystic Fibrosis Questionnaire-Revised. Value Health. 2023 Apr;26(4):567-578. doi: 10.1016/j.jval.2022.12.002. Epub 2022 Dec 9. PMID 36509366
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662
- [Derived] Rowe SM, Daines C, Ringshausen FC, Kerem E, Wilson J, Tullis E, Nair N, Simard C, Han L, Ingenito EP, McKee C, Lekstrom-Himes J, Davies JC. Tezacaftor-Ivacaftor in Residual-Function Heterozygotes with Cystic Fibrosis. N Engl J Med. 2017 Nov 23;377(21):2024-2035. doi: 10.1056/NEJMoa1709847. Epub 2017 Nov 3. PMID 29099333

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 248 participants were enrolled. Out of which, 246 received at least 1 dose of study drug were included in safety set and 244 participants who carried intended cystic fibrosis transmembrane conductance regulator (CFTR) mutations were included in Full analysis set.
Pre-assignment Details: Participants were randomized to 1 of 6 treatment sequences, each of which included 2 treatment periods and 2 of 3 potential treatments (placebo, VX-661/ivacaftor [IVA], IVA). Treatment periods were separated by an 8 week wash-out period.
Groups:
- First VX-661/IVA, Then IVA: VX-661 100 milligram (mg) plus IVA 150 mg fixed dose combination (FDC) tablet and placebo matched to IVA in the morning, IVA 150 mg tablet in the evening for 8 weeks in treatment period 1 followed by IVA 150 mg tablet and placebo matched to VX-661 plus IVA FDC tablet in the morning, IVA 150 mg tablet in the evening for 8 weeks in treatment period 2. Each treatment period was separated by a minimum 8 weeks of washout period.
- First VX-661/IVA, Then Placebo: VX-661 100 mg plus IVA 150 mg FDC tablet and placebo matched to IVA in the morning, IVA 150 mg tablet in the evening for 8 weeks in treatment period 1 followed by placebo matched to VX-661 plus IVA FDC tablet and placebo matched to IVA tablet in the morning, placebo matched to IVA tablet in the evening for 8 weeks in treatment period 2. Each treatment period was separated by a minimum 8 weeks of washout period.
- First IVA, Then Placebo: IVA 150 mg tablet and placebo matched to VX-661 plus IVA FDC tablet in the morning, IVA 150 mg tablet in the evening for 8 weeks in treatment period 1 followed by placebo matched to VX-661 plus IVA FDC tablet and placebo matched to IVA tablet in the morning, placebo matched to IVA tablet in the evening for 8 weeks in treatment period 2. Each treatment period was separated by a minimum 8 weeks of washout period.
- First IVA, Then VX- 661/IVA: IVA 150 mg tablet and placebo matched to VX-661 plus IVA FDC tablet in the morning, IVA 150 mg tablet in the evening for 8 weeks in treatment period 1 followed by VX-661 100 mg plus IVA 150 mg FDC tablet and placebo matched to IVA tablet in the morning, IVA 150 mg tablet in the evening for 8 weeks in treatment period 2. Each treatment period was separated by a minimum 8 weeks of washout period.
- First Placebo, Then VX- 661/IVA: Placebo matched to VX-661 plus IVA FDC tablet and placebo matched to IVA tablet in the morning, placebo matched to IVA tablet in the evening for 8 weeks in treatment period 1 followed by VX-661 100 mg plus IVA 150 mg FDC tablet and placebo matched to IVA tablet in the morning, IVA 150 mg tablet in the evening for 8 weeks in treatment period 2. Each treatment period was separated by a minimum 8 weeks of washout period.
- First Placebo, Then IVA: Placebo matched to VX-661 plus IVA FDC tablet and placebo matched to IVA tablet in the morning, placebo matched to IVA tablet in the evening for 8 weeks in treatment period 1 followed by IVA 150 mg tablet and placebo matched to VX-661 plus IVA FDC tablet in the morning, IVA 150 mg tablet in the evening for 8 weeks in treatment period 2. Each treatment period was separated by a minimum 8 weeks of washout period.
Period: Treatment Period 1 (8 Weeks)
Arm/Group | First VX-661/IVA, Then IVA | First VX-661/IVA, Then Placebo | First IVA, Then Placebo | First IVA, Then VX- 661/IVA | First Placebo, Then VX- 661/IVA | First Placebo, Then IVA
Started | 41 | 43 | 40 | 42 | 41 | 41
Treated | 41 | 43 | 39 | 42 | 40 | 41
Completed | 38 | 43 | 38 | 41 | 37 | 38
Not Completed | 3 | 0 | 2 | 1 | 4 | 3
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Pregnancy | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Noncompliance | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized but not treated | 0 | 0 | 1 | 0 | 1 | 0
Period: Treatment Period 2 (8 Weeks)
Arm/Group | First VX-661/IVA, Then IVA | First VX-661/IVA, Then Placebo | First IVA, Then Placebo | First IVA, Then VX- 661/IVA | First Placebo, Then VX- 661/IVA | First Placebo, Then IVA
Started | 38 | 43 | 38 | 41 | 37 | 38
Completed | 37 | 43 | 38 | 41 | 37 | 38
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) was defined as all randomized subjects who carry the intended cystic fibrosis transmembrane conductance regulator (CFTR) mutations and had received at least 1 dose of study drug.
Groups:
- First VX- 661/IVA, Then IVA: VX-661 100 mg plus IVA 150 mg FDC tablet and placebo matched to IVA in the morning, IVA 150 mg tablet in the evening for 8 weeks in treatment period 1 followed by IVA 150 mg tablet and placebo matched to VX-661 plus IVA FDC tablet in the morning, IVA 150 mg tablet in the evening for 8 weeks in treatment period 2. Each treatment period was separated by a minimum 8 weeks of washout period.
- Total: Total of all reporting groups
Arm/Group | First VX- 661/IVA, Then IVA | First VX-661/IVA, Then Placebo | First IVA, Then Placebo | First IVA, Then VX- 661/IVA | First Placebo, Then VX- 661/IVA | First Placebo, Then IVA | Total
Number analyzed (Participants) | 41 | 43 | 40 | 42 | 41 | 41 | 248
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 6 | 7 | 5 | 5 | 6 | 34
  Between 18 and 65 years | 36 | 37 | 33 | 37 | 34 | 35 | 212
  >=65 years | 0 | 0 | 0 | 0 | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 19 | 21 | 23 | 23 | 134
  Male | 18 | 18 | 21 | 21 | 18 | 18 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 3 | 2 | 2 | 9
  Not Hispanic or Latino | 40 | 43 | 39 | 39 | 37 | 39 | 237
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 0 | 0 | 1 | 3
  White | 39 | 42 | 40 | 42 | 39 | 39 | 241
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Study Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) at Average of Week 4 and Week 8
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: Baseline, Week 4 and Week 8 of each treatment period
Population: Full Analysis Set (FAS) included all randomized participants who carry the protocol specified cystic fibrosis transmembrane conductance regulator gene (CFTR) mutations and had received at least 1 dose of study drug. Here 'Overall Number of participants analyzed' signifies those participants who had evaluable data for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of predicted FEV1
Groups:
- Placebo: Placebo matched to VX-661/Ivacaftor (IVA) fixed dose combination (FDC) tablet and placebo matched to IVA tablet in the morning, placebo matched to IVA tablet in the evening for 8 weeks in treatment period 1 and 2.
- Ivacaftor: IVA 150 milligram (mg) tablet and placebo matched to VX-661/IVA FDC tablet in the morning, IVA 150 mg tablet in the evening for 8 weeks in treatment period 1 and 2.
- VX-661/IVA: VX-661 100 mg/IVA 150 mg FDC tablet and placebo matched to IVA in the morning, IVA 150 mg tablet in the evening for 8 weeks in treatment period 1 and 2.
Arm/Group | Placebo | Ivacaftor | VX-661/IVA
Number analyzed (Participants) | 160 | 156 | 159
percentage of predicted FEV1 | -0.3 [-1.2 to 0.6] | 4.4 [3.5 to 5.3] | 6.5 [5.6 to 7.3]
Statistical Analysis 1: Comparison: Placebo vs Ivacaftor; Test type: Superiority; p < 0.0001, Linear Mixed Effects Model; Least Squares (LS) Mean Difference = 4.7, 95% CI 2-sided [3.7 to 5.8]
Statistical Analysis 2: Comparison: Placebo vs VX-661/IVA; Test type: Superiority; p < 0.0001, Linear Mixed Effects Model; LS Mean Difference = 6.8, 95% CI 2-sided [5.7 to 7.8]

2. Secondary Outcome: Absolute Change From Study Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score at Average of Week 4 and Week 8
Description: The CFQ-R assessed respiratory symptoms on a scale with scores ranging from 0 to 100; where higher scores indicated fewer symptoms and better health-related quality of life.
Time Frame: Baseline, Week 4 and Week 8 of each treatment period
Population: FAS was used. Here 'Overall Number of participants analyzed' signifies those participants who had evaluable data for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- VX-661/IVA: IVA 150 milligram (mg) tablet and placebo matched to VX-661/IVA FDC tablet in the morning, IVA 150 mg tablet in the evening for 8 weeks in treatment period 1 and 2.
Arm/Group | Placebo | Ivacaftor | VX-661/IVA
Number analyzed (Participants) | 160 | 156 | 161
units on a scale | -1.0 [-2.9 to 1.0] | 8.7 [6.8 to 10.7] | 10.1 [8.2 to 12.1]
Statistical Analysis 1: Comparison: Placebo vs Ivacaftor; Test type: Superiority; p < 0.0001, Linear Mixed Effects Model; LS Mean Difference = 9.7, 95% CI 2-sided [7.2 to 12.2]
Statistical Analysis 2: Comparison: Placebo vs VX-661/IVA; Test type: Superiority; p < 0.0001, Linear Mixed Effects Model; LS Mean Difference = 11.1, 95% CI 2-sided [8.7 to 13.6]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 28
Population: Safety Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | Ivacaftor | VX-661/IVA
Number analyzed (Participants) | 162 | 157 | 162
participants
  Participants with any AEs | 126 | 114 | 117
  Participants with SAEs | 14 | 10 | 8

4. Secondary Outcome: Relative Change From Study Baseline in ppFEV1 at Average of Week 4 and Week 8
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: Baseline, Week 4 and Week 8 of each treatment period
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Ivacaftor | VX-661/IVA
Number analyzed (Participants) | 160 | 156 | 159
percent change | -0.2 [-1.7 to 1.4] | 7.9 [6.4 to 9.4] | 11.2 [9.7 to 12.7]
Statistical Analysis 1: Comparison: Placebo vs Ivacaftor; Test type: Superiority; p < 0.0001, Linear Mixed Effects Model; LS Mean Difference = 8.1, 95% CI 2-sided [6.3 to 9.9]
Statistical Analysis 2: Comparison: Placebo vs VX-661/IVA; Test type: Superiority; p < 0.0001, Linear Mixed Effects Model; LS Mean Difference = 11.4, 95% CI 2-sided [9.6 to 13.2]

5. Secondary Outcome: Absolute Change From Study Baseline in Sweat Chloride at Average of Week 4 and Week 8
Time Frame: Baseline, Week 4 and Week 8 of each treatment period
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: millimoles per liter (mmol/L)
Arm/Group | Placebo | Ivacaftor | VX-661/IVA
Number analyzed (Participants) | 151 | 153 | 151
millimoles per liter (mmol/L) | -0.4 [-2.3 to 1.5] | -4.9 [-6.7 to -3.0] | -9.9 [-11.8 to -8.0]
Statistical Analysis 1: Comparison: Placebo vs Ivacaftor; Test type: Superiority; p < 0.0001, Linear Mixed Effects Model; LS Mean Difference = -4.5, 95% CI 2-sided [-6.7 to -2.3]
Statistical Analysis 2: Comparison: Placebo vs VX-661/IVA; Test type: Superiority; p < 0.0001, Linear Mixed Effects Model; LS Mean Difference = -9.5, 95% CI 2-sided [-11.7 to -7.3]

6. Secondary Outcome: Trough Plasma Concentrations (Ctrough) of VX-661, VX-661 Metabolites (M1 VX-661), IVA and IVA Metabolite (M1 IVA) After Administration of VX-661/IVA Combination Therapy
Time Frame: Pre-morning dose on Week 8 of each treatment period
Population: Pharmacokinetic (PK) set included all randomized participants who received any amount of study drug and had a PK assessment.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | VX-661/IVA
Number analyzed (Participants) | 161
nanogram per milliliter (ng/mL)
  VX-661 | 2370 (1330)
  M1 VX-661 | 5230 (1940)
  IVA: number analyzed (Participants) | 157
  IVA | 909 (530)
  M1 IVA: number analyzed (Participants) | 159
  M1 IVA | 2010 (1050)

7. Secondary Outcome: Ctrough of IVA and IVA Metabolite (M1 IVA) After Administration of IVA Monotherapy
Time Frame: Pre-morning dose on Week 8 of each treatment period
Population: PK set was used. Here 'Overall Number of participants analyzed' signifies those participants who had evaluable data for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ivacaftor
Number analyzed (Participants) | 155
ng/mL
  IVA: number analyzed (Participants) | 154
  IVA | 696 (435)
  M1 IVA | 1550 (808)

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 28
Arm/Group | Placebo | Ivacaftor | VX-661/IVA
All-Cause Mortality (participants affected / at risk) | 0/162 | 0/157 | 0/162
Serious Adverse Events (participants affected / at risk) | 14/162 | 10/157 | 8/162
Other Adverse Events (participants affected / at risk) | 87/162 | 54/157 | 80/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=162) | Ivacaftor (N=157) | VX-661/IVA (N=162)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 8 | 6 | 4
Influenza (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 0
Pulmonary function test decreased (Investigations) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=162) | Ivacaftor (N=157) | VX-661/IVA (N=162)
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 17 | 23
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 11 | 12 | 14
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 12 | 17 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 3 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 7 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 6
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 25 | 14 | 19
Nasopharyngitis (Infections and infestations) | 5 | 6 | 13
Diarrhoea (Gastrointestinal disorders) | 10 | 5 | 13
Nausea (Gastrointestinal disorders) | 10 | 3 | 9
Headache (Nervous system disorders) | 13 | 11 | 18
Fatigue (General disorders) | 16 | 7 | 12
Pyrexia (General disorders) | 12 | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.

DOCUMENTS (2):
  • Study Protocol (2016-06-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT02392234/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/34/NCT02392234/SAP_001.pdf